CLINICAL TRIAL: NCT04695314
Title: Effect of Foot Reflexology on Intraocular Pressure in Ocular Hypertensive and Glaucoma Patients
Brief Title: Foot Reflexology in Ocular Hypertensive and Glaucoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 24685
Record Dates: First submitted 2020-12-23; First posted 2021-01-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Ocular Hypertension; Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma | interventions — Massage

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Glaucoma Group (Experimental): Patients with glaucoma come in and get an intraocular pressure check at baseline. They get a 5 minute foot massage and then have their intraocular pressure checked every 30 minutes over 2 hour span.
  Interventions: Device: Massage
- Ocular Hypertension Group A (Experimental): Patients with OHTN come in and get an IOP check at baseline. They get a 5 minute foot massage and then have their IOP checked every 30 minutes over 2 hour span.
  2 week washout period and then patients return. Patients come in the morning to have their IOP checked. Received raised experimental shoe insert. Patients come back in the afternoon to have their IOP checked again.
  2 week washout period and then patients return. Patients come in the morning to have their IOP checked. Received sham flat shoe insert. Patients come back in the afternoon to have their IOP checked again.
  Interventions: Procedure: Experimental insert; Procedure: Sham insert
- Ocular Hypertension Group B (Active Comparator): Patients with OHTN come in and get an IOP check at baseline. They get a 5 minute foot massage and then have their IOP checked every 30 minutes over 2 hour span.
  2 week washout period and then patients return. Patients come in the morning to have their IOP checked. Received sham flat shoe insert. Patients come back in the afternoon to have their IOP checked again.
  2 week washout period and then patients return. Patients come in the morning to have their IOP checked. Received raised experimental shoe insert. Patients come back in the afternoon to have their IOP checked again.
  Interventions: Procedure: Experimental insert; Procedure: Sham insert

INTERVENTIONS:
Device: Massage — Foot reflexology board (JAPAN TSUBO HH-700) with massage focused at the base of the second and third toes
  Other Names: JAPAN TSUBO HH-700
  Arms: Glaucoma Group
Procedure: Experimental insert — Raised shoe insert, insert used for massage
  Arms: Ocular Hypertension Group A; Ocular Hypertension Group B
Procedure: Sham insert — Flat shoe insert, insert used for massage
  Arms: Ocular Hypertension Group A; Ocular Hypertension Group B

SUMMARY:
To determine the effect of foot reflexology in primary open angle glaucoma (POAG) patients and the effect of a shoe insert to perform continuous foot reflexology in ocular hypertensive (OHTN) patients.

DETAILED DESCRIPTION:
This is a prospective pilot study in glaucoma patients and a prospective therapeutic trial in ocular hypertensive patients. Patients were recruited from the Temple Ophthalmology outpatient clinic. Primary open-angle glaucoma patients were recruited from those about to have SLT for additional intraocular pressure (IOP) lowering. OHTN patients were recruited from the clinic. The glaucoma patients performed a 5-minute foot massage on a foot massage board and the IOP was checked pre-massage, post-massage and 30, 60, 90 and 120 min post massage. OHTN patients underwent a one-month drop washout and then performed a 5-minute massage using a 3D-printed shoe insert with the identical pressure checks. They then were randomly assigned to wear the shoe insert or a sham insert for one day. IOP was checked before inserting the insert and at the end of the day. The number of steps was recorded each day.

ELIGIBILITY:
The inclusion criteria for this study in each study group are as follows.

* Patients with ocular hypertension (age 30-90) who may or may not have been included in the original pilot study.
* Patients with POAG (age 30-90) who are being asked to increase therapy to further lower their IOP.

The exclusion criteria for BOTH study groups will be:

* Current participation in FR or other complementary and alternative medicine techniques who will not participate in a washout period.
* Ocular hypotensive drop treatments for ocular-hypertension who will not participate in a washout period.
* Previous eye surgery or laser treatment.
* Physical inability to perform the tasks.

Additional exclusion criteria for the Foot Insert ONLY will be:

* Diabetes
* Parkinson's Disease
* Neuropathy
* Gait Abnormalities

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure Changes in Glaucoma Patients | Collect pressure readings for baseline, after 5 minutes of massage, and every 30 minutes for 2 hours
  Glaucoma Patients
Intraocular Pressure Changes in Ocular Hypertensive Patients | Collect pressure readings for baseline, after 5 minutes of massage, and every 30 minutes for 2 hours
  Ocular Hypertensive Patients
Intraocular Pressure Changes in Ocular Hypertensive Patients | Baseline and after experimental foot insert intervention, over an average of 8 hours
  Ocular Hypertensive Patients
Intraocular Pressure Changes in Ocular Hypertensive Patients | Baseline and after sham foot insert intervention, over an average of 8 hours
  Ocular Hypertensive Patients

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University Hospital Ophthalmology Clinic, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No